



## PARTICIPANT CONSENT FORM

Title of Study: The effectiveness of group Cognitive-Behavior-Therapy (CBT) and exercise in management of depression: A three-arm randomized controlled pilot trial

Principal Investigator(s): Dr. Vincent Agyapong Phone Number(s): 780-215-7771

| | <u>Yes</u> | <u>No</u> |
|---|---|---|
| Do you understand that you have been asked to be in a research study? | | |
| Have you received and read a copy of the attached Information Leaflet? | | |
| Do you understand the benefits and risks involved in taking part in this study? | | |
| Have you had an opportunity to ask questions and discuss this study? | | |
| Do you understand that you are free to leave the study at any time, without having to give a reason and without affecting your future medical care? | | |
| Has the issue of confidentiality been explained to you? | | |
| Do you understand who will have access to your records, including personally identifiable health information? | | |
| Do you understand that the study team will access and review your medical records from 6 months prior to 6 months after your enrolment in study for study purposes? | | |
| Do you understand that the study findings will be published without any individual identifiable information? | | |
| Who explained the study to you? | | |
| I agree to take part in this study: | | |
| Signature of Research Participant | | |
| (Printed Name) Date: | | |
| Signature of witness: | | |
| I believe that the person signing this form understands what is involved in the study a agrees to participate. | and volu | ntarily |
| Signature of Investigator or Designee Date | ate | |
| THE INFORMATION SHEET MUST BE ATTACHED TO THIS CONSENT FORM AND A SIGNED | | |

Ethics ID: Pro00080975 Version: 2019-March-26